CLINICAL TRIAL: NCT00893152
Title: Perspectives on Enhancing Family Involvement in Treatment for PTSD
Brief Title: Family Involvement in Treatment for PTSD
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: DHI 08-097; CAVHS 0156_2008I (Other: CAVHS IRB)
Record Dates: First submitted 2009-05-01; First posted 2009-05-05 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Male veterans (focus groups and individual interviews)
- Group 2: Female veterans (focus groups and individual interviews)
- Group 3: Family members of participating veterans (focus groups and individual interviews)

SUMMARY:
Post-traumatic stress disorder (PTSD), prevalent among returning OEF/OIF/OND Veterans, has a powerful impact on family functioning. Good family relationships appear to moderate its impact; stressful relationships may reduce the benefits of treatment. A program that assists both Veteran and family in coping with the Veteran's PTSD could directly improve the Veteran's re-adjustment and well-being and indirectly improve his/her social and occupational functioning.

DETAILED DESCRIPTION:
Background: Post-traumatic stress disorder (PTSD), a potentially severe and persistent condition that affects social, occupational and family functioning, is prevalent among returning OIF/OEF veterans. PTSD has a powerful impact on family functioning. Because good family relationships appear to moderate its impact, while stressful relationships may reduce the benefits of treatment, a program that enhances family functioning by assisting both veteran and family in coping with the veteran's PTSD could directly improve the veteran's adjustment and well-being, and indirectly improve his/her social and occupational functioning. Effective programs for OIF/OEF veterans are urgently needed. This study will address critical gaps in knowledge about relevant needs and preferences of OIF/OEF veterans and families, and how best to involve families in treatment.

Objectives: The specific aim of this project is to describe the needs and preferences of OIF/OEF service-era veterans with PTSD and their families relevant to family involvement in care.

Methods: This two-site study was conducted at the Central Arkansas Veterans Healthcare System (CAVHS, Little Rock, AR) and Oklahoma City (OKC) VAMCs. Qualitative (focus-group or individual) interviews were conducted with 47 Veterans (33 CAVHS, 14 OKC) and 36 Veteran-designated family members (19 CAVHS/17 OKC). Veterans were eligible if they were 18-65 years of age, had served in Iraq or Afghanistan since October 2001, had received treatment for PTSD at the CAVHS or OKC VAMCs in the previous 12 months, and had an adult family member who might be willing to participate in an interview. Family was defined broadly to include relatives, significant others, and friends the Veteran considered "as close as family." Interviews addressed perceived needs related to the Veteran's readjustment to civilian life, desires for family involvement in treatment, types of services that were/would have been helpful and attractive during readjustment, as well as logistic considerations (e.g., frequency of meetings). Qualitative data were analyzed using the techniques of constant comparison and content analysis. Demographic data, deployment data, and data on preferred program structure and format were collected via an anonymous paper-and-pencil questionnaire administered following the qualitative interview.

Status: Data collection and analysis of main themes are complete. In depth analysis of additional themes is ongoing.

ELIGIBILITY:
Inclusion Criteria:

Veteran:

1. Age 18-65;
2. 2 or more inpatient or outpatient mental health contacts at LR or OKC VAMC in the previous 12 months with a primary diagnosis of PTSD;
3. Served in Iraq or Afghanistan since 10/7/01;
4. Have a family member who may be willing to participate in the focus group.

Family:

1. Age > 18
2. English speaking
3. Be the designated "family member" of a participating veteran

Exclusion Criteria:

* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veteran participants were OIF/OEF veterans receiving outpatient treatment for PTSD at the Little Rock or Oklahoma City VAMCs. Each veteran participant was asked to designate an adult family member/friend to participate in a separate interview.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen P. Fischer, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System (North Little Rock)
Locations (2):
- United States (2):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas
  - VA Medical Center, Oklahoma City, Oklahoma City, Oklahoma

RESULTS

PARTICIPANT FLOW:
Groups:
- Veterans: Participants in focus groups or individual qualitative interviews
- Family Members: Family members of participating veterans who also took part in a focus group or individual qualitative interview
Period: Overall Study
Arm/Group | Veterans | Family Members
Started | 47 | 36
Completed | 47 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Veterans | Family Members | Total
Number analyzed (Participants) | 47 | 36 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (10.9) | 39.1 (13.1) | 38.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 27 | 43
  Male | 31 | 9 | 40
Region of Enrollment [Number; unit: participants]
  United States | 47 | 36 | 83

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Interviews - Perspectives on Family Involvement in PTSD Treatment
Description: This is qualitative research. "Outcomes" were themes raised with regard to content to be included in a multi-family group psychoeducation program for OEF/OIF/OND veterans with PTSD and family members.
Time Frame: During the 1-1.5 hour interviews
Population: Participants in focus group or individual qualitative interviews
Measure: Number; unit: participants
Arm/Group | Veterans | Family Members
Number analyzed (Participants) | 47 | 36
participants
  Information on Services & PTSD | 33 | 20
  Skills Training | 27 | 16
  Emotional & Instrumental Support | 12 | 17
  Perspective on the Other's Experience | 19 | 5
Statistical Analysis 1: Comparison: Veterans vs Family Members; Test type: Superiority or Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 22 months.
Description: Duration of data collection (one-time qualitative interview).
Arm/Group | Veterans | Family Members
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/36
Other Adverse Events (participants affected / at risk) | 0/47 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes